CLINICAL TRIAL: NCT02237690
Title: A Randomized, Open Label, Single-Dose, Two-Cycle Crossover Study to Assess Bioequivalence of Test and Reference Formulations of Doxorubicin Hydrochloride Liposome Injection in Female Patients With Ovarian Cancer
Brief Title: Assess Bioequivalence of Two Formulations of Doxorubicin Hydrochloride Liposome in Female Patients With Ovarian Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai Fudan-Zhangjiang Bio-Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: Libaoduo-BE-002
Record Dates: First submitted 2014-08-31; First posted 2014-09-11 (Estimated); Last update posted 2017-06-05 (Actual); Status verified 2017-06

CONDITIONS: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- doxorubicin hydrochloride liposome（Libaoduo） (Experimental): Use the test drug(doxorubicin hydrochloride liposome-Libaoduo,from Fudan-Zhangjiang ),then use the reference drug(doxorubicin hydrochloride liposome，from Sunpharma) after at least 4-weeks.
  Interventions: Drug: Doxorubicin hydrochloride liposome
- doxorubicin hydrochloride liposome (Active Comparator): Use the reference drug(doxorubicin hydrochloride liposome，from Sunpharma),then use the test drug drug(doxorubicin hydrochloride liposome-Libaoduo,from Fudan-Zhangjiang) after at least 4-weeks.
  Interventions: Drug: Doxorubicin hydrochloride liposome

INTERVENTIONS:
Drug: Doxorubicin hydrochloride liposome — 50mg/m2,IV on day1 of each cycle,On Day 1 of Cycle 2, patients will crossover to the alternate reference or test formulation,After completion of Cycle 2 (Day 28), patients will be continued on the treatment of Doxorubicin Hydrochloride Liposome Injection up to 4 more cycles if tolerance permits under guidance of their attending physicians.

SUMMARY:
This is a multi-center, single-dose, open-label, randomized, balanced, two-treatment, two-cycle, two-sequence crossover study to assess bioequivalence of test (T) and reference (R) formulations of doxorubicin hydrochloride liposome injection in female patients with ovarian cancer.

Each patient will be randomized to one of two treatment sequences (RT or TR) according to a randomization scheme prepared prior to the start of the trial.There will be at least 4-week apart between each single-dose administration. Serial blood samples for determination of free doxorubicin and liposomal encapsulated doxorubicin plasma concentrations for PK analysis will be obtained in each cycle.

The 90% confidence intervals on the GMR(geometric mean ratio) of test to reference products of free and liposome encapsulated doxorubicin for PK must be within 80-125% to demonstrate bioequivalence.

DETAILED DESCRIPTION:
This study has an adaptive 2-stage design. Bioequivalence based on encapsulated doxorubicin will be tested at the end of Stage 1 . An interim analysis of free doxorubicin will be performed at the end of Stage 1 . If needed, the study may continue into Stage 2 with additional number of ovarian cancer patients determined based on the interim analysis; and a final evaluation of bioequivalence for free doxorubicin will be performed at the end of Stage 2. Each patient will be randomized to one of two treatment sequences (RT or TR) according to a randomization scheme prepared prior to the start of the trial. Serial blood samples for determination of free doxorubicin and liposomal encapsulated doxorubicin plasma concentrations for PK analysis will be obtained in each cycle.

The 90% confidence intervals on the GMR（geometric mean ratio） of test to reference products of free and liposome encapsulated doxorubicin for PK must be within 80-125% to demonstrate bioequivalence.

Safety data will be summarized and listed. Adverse events will be coded and classified by system organ class and preferred term using Common Terminology Criteria for Adverse Events. A summary of all drug-related adverse events will also be generated. Clinical laboratory data will be summarized descriptively and listed by treatment group. The change from pre dose to the end of the study will also be summarized. Prior and concomitant medications will be coded with the World Health Organization Drug Dictionary and listed. Vital signs and electrocardiogram data will be summarized and listed by dose group and visit.

ELIGIBILITY:
Inclusion Criteria:

* Able to give written informed consent for participation in the trial;
* Females age 18 to 75 years, inclusive;
* Histologically or cytologically proven ovarian cancer, which has progressed or recurred by CT/MRI confirmation after platinum-based chemotherapy;
* ECOG (Eastern Cooperative Oncology Group) Performance Status 0 - 2;
* Patient is expected to be able to receive both doses of Doxorubicin Hydrochloride Liposome Injection and participate in the trial for at least 56 days.
* Urine pregnancy test before dosing of both cycle1 and cycle 2 must be negative (not including postmenopausal or surgically sterile women); Agree to use an approved method of birth control (condom with spermicide, diaphragm or cervical cap with spermicide, or intrauterine device); or patients of non-childbearing potential who are either surgically sterile (hysterectomy, bilateral oophorectomy, or bilateral tubal ligation) or >1 year postmenopausal with follicle-stimulating hormone in the postmenopausal range;

  * 30days or 5 half-lives (whichever is longer) have elapsed from the completion of previous cancer therapy, and patients must have recovered to < Grade 2 or be at new stable baseline from any related toxicities;
* Adequate renal, hepatic and bone marrow function without blood product or hematopoietic growth factor support:
* Able to comply with study requirements in the opinion of the Principal Investigator

Exclusion Criteria:

* Significant allergy, hypersensitivity or idiosyncratic reactions to doxorubicin and/or any related compounds;
* History or presence of cardiac disease rated New York State Heart Association Classification class 2 or greater;
* Uncontrolled cardiac arrhythmia or other findings on screening electrocardiogram (ECG) which could, in the judgment of the Principal Investigator, put the patient at undue risk for participation in the trial;
* LVEF（left ventricular ejection fraction） below 50% or below institutional normal at screening;
* Prior radiation therapy to mediastinum;
* Concomitant use of other cytotoxic or cytostatic drugs or of radiotherapy;
* Active, uncontrolled infection, including opportunistic infection with mycobacteria, cytomegalovirus, toxoplasma, or P. carinii;
* Use of prescription or non-prescription herbal and dietary supplements, within 7 days or 5 half-lives (whichever is longer) prior to the first dose of study medication.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2015-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
pharmacokinetic（PK） parameter:the maximum plasma doxorubicin concentrations(Cmax) | 2 cycles
  The study endpoint will use the PK parameter(Cmax) for free doxorubicin and liposome encapsulated doxorubicin
PK parameter:the areas under the plasma concentration versus time curve calculated from 0 to the last measurable observation(AUC0-t) | 2 cycles
  The study endpoint will use the PK parameter(AUC0-t) for free doxorubicin and liposome encapsulated doxorubicin(AUC0-t)
PK parameter:the areas under the plasma concentration versus time curve extrapolated from 0 to infinity(AUC0-inf) | 2 cycles
  The study endpoint will use the PK parameter(AUC0-inf) for free doxorubicin and liposome encapsulated doxorubicin

SECONDARY OUTCOMES:
incidence of treatment-emergent adverse events (TEAEs) | 2 cycles
study discontinuation information | 2 cycles

CONTACTS AND LOCATIONS:
Overall Officials: Wu li ngying, Ph.D, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences; Kong be ihua, Ph.D, Principal Investigator — Shandong University Qilu Hospital; Liu ji hong, Ph.D, Principal Investigator — Sun Yat-sen University
Locations (3):
- China (3):
  - Cancer Institute& Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - QiLu Hospital of Shandong University, Jinan, Shandong